CLINICAL TRIAL: NCT03416517
Title: Anlotinib and Irinotecan for Advanced Ewing Sarcoma After Failure of Standard Multimodal Therapy
Brief Title: Anlotinib and Irinotecan for Ewing Sarcoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, GUO WEI, Director of Musculoskeletal Tumor Center, Peking University People's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-EWS-02
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Ewing's Tumor Metastatic
Keywords: Ewing Sarcoma; Anlotinib; Irinotecan; Refractory; Metastatic
MeSH Terms: conditions — Sarcoma, Ewing; Neoplasm Metastasis | interventions — anlotinib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib and Irinotecan(phase 1b) (Experimental): Anlotinib 12 or 8 mg/d PO on days 1-14 q3w. Irinotecan 20 or 15mg/m^2/d over 60 minutes on days 1-5 and 8-12 q3w. Vincristine 1.4mg/m^2/d IV on days 1,8 q3w. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anlotinib; Drug: Irinotecan
- Anlotinib and Irinotecan(phase 2) (Experimental): Anlotinib 12 or 8 mg/d PO on days 1-14 q3w. Irinotecan 20 or 15 mg/m^2/d IV over 60 minutes on days 1-5 and 8-12 q3w. The final dose of anlotinib and irinotecan depends on the result from previous phase Ib study. Vincristine 1.4mg/m^2/d IV on days 1,8 q3w. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anlotinib; Drug: Irinotecan

INTERVENTIONS:
Drug: Anlotinib — Anlotinib 12 or 8 mg/d po D1-14 q3w
  Other Names: AL3818
Drug: Irinotecan — Irinotecan 20 or 15mg/m^2/d IV over 60 minutes on days 1-5 and 8-12, q3w
  Other Names: Camptosar

SUMMARY:
The investigators explored the activity of anlotinib combined with irinotecan in patients with relapsed and metastatic Ewing Sarcoma.

DETAILED DESCRIPTION:
After standard multimodal therapy, the prognosis of relapsed and metastatic Ewing Sarcoma is dismal and unchanged over the last decades.Thus, the investigators explored the activity of anlotinib combined with irinotecan in patients with relapsed and metastatic Ewing Sarcoma after the failure of first-line chemotherapy with doxorubicin, vincristine, cyclophosphamide, ifosphamide and etoposide.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Ewing sarcoma.
* Evidence of Ewing sarcoma translocation by fluorescence in situ hybridization (FISH) or real-time polymerase chain reaction (RT-PCT).
* Recurrent or refractory tumors with no known curative treatment options according to the judgment of the investigator.
* Prior treatment consisted of standard Ewing Sarcoma chemotherapy agents including doxorubicin, vincristine, cyclophosphamide, ifosfamide and etoposide; metastatic relapsed and unresectable progressive disease (PD);
* Life expectancy of ≥ 3 months.
* Eastern Cooperative Oncology Group performance status 0-1
* Measurable disease on CT or MRI by RECIST 1.1.
* Adequate organ function.
* Time elapsed from previous therapy must be ≥ 3 weeks for systemic therapy, ≥ 2 weeks for radiation therapy or major surgery.
* Patients who have undergone autologous hematopoietic stem cell transplantation are eligible once they have recovered from all toxicities from therapy.
* Patients who have received allogeneic hematopoietic stem cell transplantation will be eligible 6 months after the procedure provided there is no evidence of active graft-versus-host disease and immunosuppressive treatment has been discontinued for at least 30 days.
* Patients with central nervous system disease are eligible for enrollment if they have received prior radiotherapy or surgery to sites of central nervous system metastatic disease, have been off glucocorticoids for at least 4 weeks, have no overt evidence of neurological deficit and are ≥ 6 weeks from completion of brain irradiation.
* Females of childbearing potential as well as males and their partners must agree to use an effective form of contraception during the study and for 6 months following the last dose of study medication.

Exclusion Criteria:

* Clinically significant unrelated illness which would, in the judgment of the treating physician, compromise the patient's ability to tolerate the investigational agent or be likely to interfere with the study procedures or results.
* Prior treatment consisted of anlotinib, any other antiangiogenic TKIs, or irinotecan.
* Patients with baseline corrected QT interval(QTc) > 480 msec.
* Known hypersensitivity reaction to anlotinib or any of its components, and irinotecan or any of its components.
* Concomitant use of any other investigational or anticancer agent(s).
* Pregnant patients or patients who are breast feeding. Subjects capable of pregnancy (post menarche and not post-menopausal, defined as over 12 months since final menstrual period) must have a negative pregnancy test within 7 days prior to first dose.
* Inability to swallow capsules or water.
* Other clinically significant malignant disease diagnosed within the previous 5 years, excluding intra-epithelial cervical neoplasia or non-melanoma skin cancer.
* Known persistent (> 4 weeks) ≥ Grade 2 neutropenia, ≥ Grade 2 thrombocytopenia or > Grade 3 anemia from prior cancer therapy.
* Other kinds of malignant tumors at the same time.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (phase 1b) | 12 months
  evaluate the maximum tolerated dose (MTD) of combination therapy with irinotecan and anlotinib
Object response rate(ORR) at 12 weeks (phase 2) | 12 months
  complete response (CR) + partial response (PR) at 12 weeks

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 2 years
  Calculated from the date of treatment start until the time of disease progression or death, whichever comes first.
Overall survival(OS) | 2 years
  Calculated from the date of treatment start until last follow-up or death, whichever comes first.
Adverse Effect | 2 years
  Adverse effect measured by CTCAE v.4 (Common Terminology Criteria for Adverse Events)
Quality of Life (QoL) | 2 years
  Quality of Life measured by EORTC QLQ(quality of life questionnair) C-30 for adults or PedsQL3.0 for children.
Pain management | 2 years
  Pain management measured by Visual Analog Score for pain.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D, Ph.D, Principal Investigator — Peking University People's Hospital
Locations (5):
- China (5):
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Shougang Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - People's Liberation Army General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dong S, Sun K, Xie L, Xu J, Sun X, Ren T, Huang Y, Yang R, Tang X, Yang F, Gu J, Guo W. Quality of life and Q-TWiST were not adversely affected in Ewing sarcoma patients treated with combined anlotinib, irinotecan, and vincristine: (Peking University People's Hospital Ewing sarcoma trial-02, PKUPH-EWS-02). Medicine (Baltimore). 2021 Dec 23;100(51):e28078. doi: 10.1097/MD.0000000000028078. PMID 34941047